CLINICAL TRIAL: NCT05420415
Title: The Tumor Microenvironment Collagen Signature (CSTME) Associates With the Prognosis of Stage II and III Colorectal Cancer : A Multi-Center Retrospective Observational Cohort Study
Brief Title: The CSTME Associates With the Prognosis of Stage II and III Colorectal Cancer
Acronym: CRC23_CSTME
Status: Completed | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC22-192
Record Dates: First submitted 2022-06-12; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — paraffin tissue section
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-CSTME: Patients with high tumor microenvironment collagen signature
  Interventions: Other: CSTME
- Low-CSTME: Patients with low tumor microenvironment collagen signature

INTERVENTIONS:
Other: CSTME — Tumor microenvironment collagen signature
  Groups: High-CSTME

SUMMARY:
Colorectal cancer (CRC) is the second most commonly occurring cancer worldwide. Thirty-five percent of CRC patients are diagnosed at stage II/III, and their outcome differs even if they are in the same stage. Previous study found that the microenvironmental collagen is associated with tumor progression and metastasis. Whether tumor microenvironmental collagen signature is associated with colorectal cancer prognosis still remains unknown. We hypothesize that the tumor microenvironmental collagen signature of colorectal cancer is associated with prognosis.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second most commonly occurring cancer worldwide. Thirty-five percent of CRC patients are diagnosed at stage II/III, and their outcome differs even if they are in the same stage. In the "seed and soil" theory proposed by Stephen Paget, tumor cells play the role of the "seed", and the tumor microenvironment (TME) is the "soil". TNM classification provides useful but uncomplete prognosis information in colorectal cancer. It lacks the assessment of the "soil" signature of tumor microenvironment. Previous study found that the microenvironmental collagen is associated with tumor progression and metastasis. Whether tumor microenvironmental collagen signature is associated with colorectal cancer prognosis still remains unknown.

This study is a retrospective observational study performed in two centers. The main purpose of this study was to investigate whether the tumor microenvironment collagen signature (CSTME) can discriminate the 5-year DFS of stage II/III CRC patients, the secondary purpose is to compare the AUC (area under the receiver operating characteristic curve) of TNM stage+CSTME in predicting 5-year DFS with that of TNM stage alone. This study would introduce the tumor microenvironmental collagen signature into current colorectal cancer classification system, which would provide reference for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed with colorectal cancer
* TNM stages II and III (according to the 8th edition of AJCC Cancer Staging Manual)
* Received radical tumor resection surgery

Exclusion Criteria:

* ASA grade 4
* Preoperative radiotherapy and/or chemotherapy
* Hereditary colorectal cancer
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with stageII/III colorectal cancer
Sampling Method: Probability Sample
Enrollment: 570 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
5-year DFS | 5 years followup after surgery
  5-year disease free survival

SECONDARY OUTCOMES:
5-year OS | 5 years followup after surgery
  5-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jun Yan, MD, Study Chair — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided